CLINICAL TRIAL: NCT02374190
Title: The Relationship Between Off-hours Admissions for Primary Percutaneous Coronary Intervention, Door-to-balloon Time and Mortality for Patients With ST-elevation Myocardial Infarction in England: a Registry-based Prospective National Cohort Study
Brief Title: Relationship Between Primary Percutaneous Coronary Intervention, Door-to-balloon Times, and Mortality for Heart Attack Patients Across England
Status: Completed | Type: Observational
Sponsor: London School of Economics and Political Science (Other)
Responsible Party: Sponsor
Other Study IDs: LSEHE40914022015
Record Dates: First submitted 2015-02-13; First posted 2015-02-27 (Estimated); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (1):
- Hospital Admitted STEMI Patients: The analytical cohort for this study consisted of STEMI patients aged over 18 years admitted directly to '24/7' PPCI-capable hospitals for PPCI. STEMI patients were identified based on their discharge diagnoses and were selected as having received PPCI according to their initial reperfusion strategy. Hospitals performing only sporadic PPCI procedures, which we defined as less than 20 procedures per year, and only performing PPCIs during regular hours were not included in the analysis. Interhospital transfers were not included in the analysis, and we limited our analysis to PPCIs conducted within 6 hours on hospital arrival on the assumption that patients with a DTB time beyond this did not receive PCI as a primary reperfusion strategy. The analysis was conducted for the time period for which data were available-1 January 2007 to 31 December 2012. We conducted a complete-case analysis.
  Interventions: Other: Standard Hospital Care

INTERVENTIONS:
Other: Standard Hospital Care — We described patient characteristics using percentages for categorical data, means and SD or medians and IQRs for normally and non-normally distributed continuous variables, respectively. Statistical comparisons for differences in baseline characteristics among patients admitted during regular hours and off-hours were performed using χ2 tests for categorical variables, t-tests and Wilcoxon rank sum tests for normally and non-normally distributed continuous variables, respectively. DTB times were described using median and IQR based on time of admission. All p values were calculated as two-tailed analyses, using a significance level of 5%.

SUMMARY:
The degree to which elevated mortality associated with weekend or night-time hospital admissions reflects poorer quality of care ('off-hours effect') is a contentious issue. We examined if off-hours admissions for primary percutaneous coronary intervention (PPCI) were associated with higher adjusted mortality and estimated the extent to which potential differences in door-to-balloon (DTB) times-a key indicator of care quality for ST elevation myocardial infarction (STEMI) patients-could explain this association. Nationwide registry-based prospective observational study using Myocardial Ischemia National Audit Project data in England. We examined how off-hours admissions and DTB times were associated with our primary outcome measure, 30-day mortality, using hierarchical logistic regression models that adjusted for STEMI patient risk factors. In-hospital mortality was assessed as a secondary outcome. Our study found that higher adjusted mortality associated with off-hours admissions for PPCI could be partly explained by differences in DTB times.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients admitted from 1 January 2007 to 31 December 2012
* STEMI patients aged over 18 years
* STEMI patients admitted directly to '24/7' PPCI-capable hospitals for PPCI
* Discharge diagnosis of STEMI
* Provision of PPCI based on initial reperfusion strategy

Exclusion Criteria:

* Hospitals performing less than 20 procedures per year
* Hospitals performing PPCIs only during regular hours
* Interhospital transfers
* PPCIs conducted within 6 hours on hospital arrival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patients admitted to hospital in England for STEMI between 1 January 2007 and 31 December 2012.
Sampling Method: Non-Probability Sample
Enrollment: 42677 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2019-12-24 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days post-discharge

SECONDARY OUTCOMES:
In-hospital mortality | Patient length of stay in hospital until discharge, an average of 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Elias Mossialos, MD PhD, Principal Investigator — London School of Economics and Political Science; Sebastian Salas-Vega, PhD, Principal Investigator — London School of Economics and Political Science; Sahan Jayawardana, MSc, Study Chair — London School of Economics and Political Science
Locations (1):
- London School of Economics and Political Science, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jayawardana S, Salas-Vega S, Cornehl F, Krumholz HM, Mossialos E. The relationship between off-hours admissions for primary percutaneous coronary intervention, door-to-balloon time and mortality for patients with ST-elevation myocardial infarction in England: a registry-based prospective national cohort study. BMJ Qual Saf. 2020 Jul;29(7):541-549. doi: 10.1136/bmjqs-2019-010067. Epub 2019 Dec 12. PMID 31831635